CLINICAL TRIAL: NCT04888728
Title: An Open Label, 2-part, One-sequence, 3-period Study to Evaluate Drug-drug Interactions Between "DWN12088" and "Nebivolol" or "Paroxetine" in Healthy Male Volunteers
Brief Title: To Evaluate Drug-drug Interactions Between DWN12088 and Nebivolol or Paroxetine in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DW_DWN12088104
Record Dates: First submitted 2021-04-28; First posted 2021-05-17 (Actual); Last update posted 2021-08-04 (Actual); Status verified 2021-08

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — Nebivolol; Paroxetine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DWN12088 and Nebivolol (Experimental): Period 1 - Nebivolol A mg, Tablet, oral, once daily, Period 2 - DWN12088 X mg, Tablet, oral, twice daily, Period 3 - 1) Nebivolol A mg, Tablet, oral, once daily & DWN12088 X mg, Tablet, oral, twice daily, 2) DWN12088 X mg, Tablet, oral, once daily
  Interventions: Drug: DWN12088; Drug: Nebivolol
- DWN12088 and Paroxetine (Experimental): Period 1 - DWN12088 X mg, Tablet, oral, once daily , Period 2 - Paroxetine B mg, Tablet, oral, once daily, Period 3 - 1) DWN12088 X mg, Tablet, oral, once daily & Paroxetine B mg, Tablet, oral, once daily, 2) Paroxetine B mg, Tablet, oral, once daily
  Interventions: Drug: DWN12088; Drug: Paroxetine

INTERVENTIONS:
Drug: DWN12088 — Prolyl-tRNA synthetase (PRS) inhibitor
Drug: Nebivolol — Nebivolol
  Arms: DWN12088 and Nebivolol
Drug: Paroxetine — Paroxetine
  Arms: DWN12088 and Paroxetine

SUMMARY:
An open label, 2-part, one-sequence, 3-period study to evaluate drug-drug interactions between DWN12088 and nebivolol or Paroxetine in healthy volunteers

ELIGIBILITY:
Inclusion Criteria:

* Healthy male adults aged ≥ 20 and ≤ 55 years at screening
* Subjects who voluntarily decided to participate in the study and provided written consent to follow study compliance requirements after receiving a detailed explanation on this study and fully understanding the information

Exclusion Criteria:

* Subjects unable to have the standard meal provided at the study site
* Subjects who took (the day of taking the last dose) another investigational or bioequivalence study product within 180 days prior to the first dose

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2021-06-30 (Actual); Primary Completion 2021-07-12 (Actual); Study Completion 2021-07-27 (Actual)

PRIMARY OUTCOMES:
Cmax of Nebivolol | Day 1, Day 2, Day 3, Day 6, Day 7, and Day 8
  Cmax of Nebivolol
AUCt of Nebivolol | Day 1, Day 2, Day 3, Day 6, Day 7, and Day 8
  AUCt of Nebivolol
Cmax of DWN12088 | Day 1, Day 2, Day 3, Day 4, Day 9, Day 10, Day 11, and Day 12
  Cmax of DWN12088
AUCt of DWN12088 | Day 1, Day 2, Day 3, Day 4, Day 9, Day 10, Day 11, and Day 12
  AUCt of DWN12088

CONTACTS AND LOCATIONS:
Overall Officials: Jong-Lyul Ghim, Principal Investigator — Busan Paik Hospital
Locations (1):
- Inje University Busan Paik Hospital, Busan, South Korea